CLINICAL TRIAL: NCT04302246
Title: Immune Functional Profile as Predictor of Infective Complications Following Pediatric Liver Transplantation
Brief Title: Immune Function Following Liver Transplantation
Acronym: SEPTIFOIE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI 11055
Record Dates: First submitted 2019-12-18; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2019-12

CONDITIONS: Liver Transplant; Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biological collection will include plasma, RNA and DNA samples, which will be stored at - 20 ° C for sera, and - 40 ° C for blood RNA and liver biopsy (stabilized in a buffer containing RNase inhibitors) and DNA (stabilized in a buffer containing DNase inhibitors)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: Biological testing on sequential blood sample — Biological characterization of various immune function and blood circulating leukocytes phenotyping before liver transplantation and therafter at day-3, -7, -14 postoperatively and if septic complication occurs.

SUMMARY:
Post-operative care following liver transplantation is characterized by a high incidence of infective and immunological complications. Restauration of liver function following liver transplantation is progressive and characterize a period of immuno-infective vulnerability. The purpose of this study is to characterize the early post-operative immune function in children after liver transplantation.

DETAILED DESCRIPTION:
Within a few decades, liver transplantation has become an effective treatment of end-stage liver diseases associated with high spontaneous mortality. However, the consequences of immediate transplants are frequently complicated by infective (nosocomial infection) and immunological complications (acute graft rejection) in up to 40 to 60% of liver transplanted patients. In order to ensure graft immunotolerance, immunosuppressive therapy based mainly on calcineurin inhibitors, is initiated soon after liver transplantation. Immunosuppressive therapy is intended to reduce the response of cytotoxic lymphocytes and NK cells. As a result, an important component of the immune response is blocked. In addition, function of the transplanted liver, which is a key organ for both immuno-inflammatory signalling and host defense against pathogens, is progressively restored post-operatively. Thus in this post-transplant period, there is a critical period where liver function is severly impaired and progressively get restaured. The aim of this study is to characterize the restauration of immune function in the early post-operative period and evaluate its correlation with occurence of infective or immunological complications.

ELIGIBILITY:
Inclusion Criteria:

* Child under 18 admitted for liver transplantation
* Signature of consent by the two holders of parental authority.
* Informing children as far as their age and condition allow.
* Affiliation to a social protection

Exclusion Criteria:

* Children under 6 kg
* Children transplanted for primary graft dysfunction
* Children scheduled for liver-kidney transplants

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Child admitted for liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-01-08; Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Immune functionnal profile | pre-operatively
  quantitative monocytes mHLA-DR measurment

CONTACTS AND LOCATIONS:
Overall Officials: Pierre TISSIERES, Principal Investigator — Assistance Publique des Hopitaux de Paris

IPD SHARING:
Plan to Share IPD: No